CLINICAL TRIAL: NCT01400438
Title: Experience of the Patient Treated With Trastuzumab (Herceptin ®) as Adjuvant for Breast Cancer: Fatigue and Quality of Life During and Waning of Treatment, Psychosocial Aspects (Environment, Work)
Brief Title: Experience of the Patient Treated With Trastuzumab (Herceptin ®) as Adjuvant for Breast Cancer
Acronym: HER-ception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: HER-ception
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: Herceptin; Breast cancer; Quality of life; fatigue
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients group with Herceptin (Experimental): Patients beginning Herceptin in adjuvant after chemotherapy
  Interventions: Other: questionnaires
- Control group (Active Comparator): patient not beginning Herceptin after chemotherapy : control group
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — delivery of questionnaires and self-psychological interview
  Arms: patients group with Herceptin
Other: questionnaires — delivery of questionnaires and self-psychological interview
  Arms: Control group

SUMMARY:
Many studies have been devoted to the quality of life of patients during adjuvant chemotherapy for breast cancer by highlighting fatigue, psychological distress and impact on the immediate environment (spouse, children) during this difficult time for women. Curiously, no study to date has been submitted or published about how women with a one-year treatment "extra" Herceptin ® live this period in terms of quality of life, in terms of psychological impact for themselves and their families.

The investigators have no more data on how often they return to work during this treatment or on the psycho-social parameters which underpin them. It therefore seemed interesting to "give a spotlight" on this particular period in these women HER2 + by comparing a patient population of same age receiving the same adjuvant but with no Herceptin ®.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 18
* Invasive breast carcinoma confirmed histologically
* Non-metastatic cancer
* Surgery of the primary tumor performed (mastectomy or lumpectomy) and associated with an audit axillary (sentinel node and / or axillary dissection)
* Patient should receive their last course of adjuvant chemotherapy (3 FEC and 3 Taxotere)
* Patients not receiving the third course of Taxotere because of toxicities may be included in the fifth course of chemotherapy is the second of Taxotere
* For the group Herceptin ®: HER2 overexpression without contraindication to treatment administration
* For the control group: no indication for Herceptin ®
* Radiation therapy and / or adjuvant hormonal therapy allowed
* Free and informed consent signed

Exclusion Criteria:

* Women under 18 or over 60 years
* Histology other than adenocarcinoma
* Metastatic Breast Cancer
* Chemotherapy neoadjuvant
* Surgery of the primary tumor unrealized
* Lack of adjuvant chemotherapy with Taxotere 3 FEC and 3
* Patients with a history of malignancy within 5 years, outside of a basal cell cancer or cancer of the cervix treated and cured
* Patient under guardianship or unable to give informed consent,
* Pregnant or lactating
* Patient unable to undergo a medical for geographical, social or psychopathological

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-07; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
score of fatigue | at 9 months
  The main objective of this study is to evaluate the score of fatigue in patients with HER2 overexpressing breast cancer and for whom Herceptin ® treatment is prescribed, compared with a population of patients treated with the same age the same chemotherapy without Herceptin ®.

SECONDARY OUTCOMES:
Assess the quality of life | 3, 6, 9 and 12 months
  Assess the quality of life of patients treated for breast cancer with surgery followed by adjuvant chemotherapy (+/-hormonotherapy) associated with treatment with Herceptin ®, compared with patients of similar age treated with the same chemotherapy without Herceptin ®
Impact of Herceptin ® in the professional lives | at 3, 6 ,9 and 12 months
  Assess the impact of Herceptin ® in the professional lives of patients, compared to patients not treated with Herceptin ®.
  Evaluation done by a specific questionnaire on professional lives, a scoring will be determined.
quantitative and qualitative psychological impact of Herceptin ® | at 3 months
  Assess the quantitative and qualitative psychological impact of Herceptin ® in patients so treated, compared to patients not treated with Herceptin ®.
  Evaluation done by specific questionnaires, a scoring will be determined.
a qualitative sociological analysis among spouses of patients | at 6 months
  Conduct a qualitative sociological analysis among spouses of patients treated with Herceptin ®.
  An interview with a sociologist will be done and characteristic sociologic of patients will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Corinne DELCAMBRE, MD, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François BACLESSE, Caen, Calvados, France